CLINICAL TRIAL: NCT06852482
Title: Simulation-based Education for Physiotherapy Facilitators and Students
Brief Title: Simulation-based Education in Physiotherapy
Acronym: SimFisio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vic - Central University of Catalonia (Other)
Responsible Party: Principal Investigator, Mirari Ochandorena Acha, Director of the Master's Degree in Physiotherapy (PhD), University of Vic - Central University of Catalonia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SimFisio01
Record Dates: First submitted 2024-12-05; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Self Efficacy; Empathy
Keywords: Simulation based education; students; facilitators; physiotherapy
MeSH Terms: interventions — Behavior Therapy

STUDY DESIGN:
Intervention Model Description: This prospective quasi-experimental study has a mixed methodological design, of an explanatory sequential type, in which two phases are differentiated: 1) in the first phase, objective 1 will be worked on and will have a quantitative design; and 2) in the second phase, objective 2 will be worked on and will have a qualitative design.
  Study population include students and facilitators in simulation-based education.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facilitator population (Other): Regarding the inclusion and exclusion criteria established for the facilitators:
  Inclusion criteria:
  a) Facilitator of simulations in the Pràcticum I, III, or V courses.
  Exclusion criteria:
  a) Failure to attend both training sessions.
  Interventions: Other: SBE Capacitation (behavioral intervention) for facilitator population
- Student population (Other): The following inclusion and exclusion criteria have been established for the student population:
  Inclusion criteria:
  1. First enrollment in the Pràcticum I, III, or V courses.
  2. Completion of the full SBE session.
  Exclusion criteria:
  a) Failure to achieve a grade of 5 in any of the evaluative components of the course.
  Interventions: Other: SBE (behavioral intervention) for student population

INTERVENTIONS:
Other: SBE Capacitation (behavioral intervention) for facilitator population — An intervention is proposed with two training sessions for the tutors of the Pràcticum I, III, and IV courses in the Physiotherapy Degree. The first session will be on January 10, 2024 (3 hours), and the second on February 2, 2024 (2 hours), both at the FCSB facilities of UVic-UCC.
  The sessions aim to:
  Promote behavior that facilitates learning in Simulation-Based Education (SBE). Provide facilitators with tools and strategies for effective SBE implementation.
  Highlight the differences and similarities in SBE across the Pràcticum I, III, and IV courses, based on increasing difficulty.
  Training will involve clinical simulation principles, with facilitators experiencing all SBE phases. An actress, later participating in student simulations, will be involved. Scenarios from the courses will be used, supported by a PowerPoint presentation and an information dossier for participants.
  Other Names: For facilitator population
  Arms: Facilitator population
Other: SBE (behavioral intervention) for student population — Simulation-Based Education Each student in Pràcticum I, III, and V will participate in a simulation session tailored to their course.
  Simulations are conducted in groups of five students with the same UVic tutor acting as facilitator. Each simulation follows three phases (prebriefing, simulation, debriefing), with varying emphasis across courses:
  Pràcticum I: The prebriefing ensures group confidence. Two volunteer students participate in the simulation. The debriefing is shorter, less focused on outcomes, and highlights learning over errors. Emphasizes guidance for student.
  Pràcticum III: Prebriefing and debriefing are equally emphasized. One volunteer student performs the simulation.
  Pràcticum V: Cases are more complex, requiring less prebriefing but comprehensive briefing. Students autonomously set session rules. The debriefing is in-depth and focuses on clinical application. One volunteer student performs the simulation, Focuses on autonomy and independent work.
  Other Names: For student population
  Arms: Student population

SUMMARY:
BACKGROUND: Simulation-based education (SBE) is a current teaching methodology characterized by providing realistic and effective environments, enhancing patient-professional clinical contact in a safe educational environment. Not all facilitators are trained to guide simulations in a systematic way. As a consequence, it is not possible to guarantee homogeneity of the methodology applied so that the simulations have better results in student learning.

OBJECTIVES: 1) To evaluate the impact of the BSE training of the Physiotherapy degree facilitators on their teaching self-efficacy; 2) To evaluate the impact of the BSE on the perceived self-efficacy, academic commitment and empathy of the 2nd, 3rd and 4th year Physiotherapy students; 3) To describe the degree of satisfaction and confidence in learning with respect to the BSE of the 2nd, 3rd and 4th year Physiotherapy students. The qualitative phase aims to know the experiences of Physiotherapy students regarding the EBS.

METHODOLOGY: Prospective quasi-experimental study of mixed methodology, in which simulation facilitators and students will be studied within the framework of the subjects Pràcticum I, III and V of the Physiotherapy degree of the FCSB. Students with a grade <5 in any of the evaluative parts of these subjects and facilitators who have not completed the two proposed training sessions will be excluded. Demographic and teaching self-efficacy variables will be collected from the facilitators at 3 points in time: before and after the training and at the end of the period of simulations of Pràcticum I, III and V.

EXPECTED BENEFITS: The present mixed methodology project is expected to bring benefits in the training of the facilitators of the EBS of the Physiotherapy degree, better methodological quality of the EBS carried out in the subjects Pràcticum I, III and V of the same degree; iii) A favorable impact on the perceived self-efficacy, academic behavior and empathy of the second, third and fourth year students of the Physiotherapy Degree; iv) To know the degree of satisfaction and confidence for learning shown by students who perform EBS in the Degree of Physiotherapy; v) To know the students' perception of the best educational practices in EBS performed in the Degree of Physiotherapy; vi) To know the experiences of the students of the Degree of Physiotherapy with respect to EBS.

DETAILED DESCRIPTION:
Clinical simulation has been shown to be a pedagogical tool that enhances students' self-confidence and facilitates the integration of fundamental practical skills acquired in the classroom, as well as "multidisciplinary skills" such as communication, collaboration and conflict resolution.

EBS can be approached using a variety of modalities, which are classified according to levels of complexity, fidelity or realism, resulting in three types: low, intermediate and high complexity. In all phases of the EBS, the facilitator guides the learner in planning (prebriefing) and conducting the simulation, establishes a safe learning environment, and facilitates reflection with debriefing.

For this reason, during the 2023-2024 academic year, training will be provided for the facilitators of the simulations in the Physiotherapy Degree, with the aim of providing tools and strategies for a more effective development of the EBS.

Methodology Study design This prospective quasi-experimental study has a mixed methodological design, of an explanatory sequential type, in which two phases are differentiated: 1) in the first phase, objective 1 will be worked on and will have a quantitative design; and 2) in the second phase, objective 2 will be worked on and will have a qualitative design. Both phases will be complementary.

Study population The study population will be the 2nd, 3rd and 4th year students of the Degree in Physiotherapy of the FCSB, who are enrolled in the subjects Practicum I, III or V of the Degree and who have received the EBS, as well as the tutors of such subjects who have a role as Facilitator in the Simulations.

Inclusion criteria: a) First enrollment in Practicum I, III or V subjects; b) Completion of the entire EBS session.

Exclusion criteria: a) Failure to obtain a grade >5 in any of the evaluative parts of the subject.

Regarding the inclusion and exclusion criteria established for the population of facilitators:

Inclusion criteria: a) Facilitator of the simulations in Practicum I, III or V subjects.

Exclusion criteria: a) Not having completed the two training sessions.

Since this is a single-group quasi-experimental study, no randomization method will be applied to the study populations.

The recruitment process for the quantitative phase will be carried out, in both populations, orally and in writing through the information and informed consent form prepared for this project.

As for the Facilitator population, the same process of explanation will be applied in a briefing session by a member of the research team and they will receive a QR code to indicate, pseudo-anonymously and privately, whether or not they decide to participate in the study.

In the qualitative phase, convenience sampling will be used on the students included in the quantitative phase and who have taken the EBS.

Data Collection During Phase 1, quantitative data will be collected using the Forms extension of Microsoft 365, via a QR code that participants will receive.

Facilitating Variables:

Independent variables:

Sociodemographic data: subject (Practicum I, III, V), age, gender, previous training in EBS. These variables will be collected at baseline.

EBS training:

An intervention is proposed in two training days for tutors of the subjects Practicum I, III and IV of the Degree in Physiotherapy. The two sessions to be held in the context of the Training will have common objectives:

To favor a facilitating behavior for learning during the application of the EBS.

To provide tools and strategies to the facilitators for the correct functioning of the EBS.

To establish the differences and similarities of the EBS between the subjects Practicum I, III and V, according to the pre-established increasing difficulty.

Dependent variables:

Debriefing for Simulation in Health (EDSS). This scale assesses facilitator behaviors that facilitate learning and change in experiential contexts, through analysis and assessment of six key elements of a debriefing.

Teaching self-efficacy by means of the Teaching Self-Efficacy Scale. The scale perceived efficacy in student and in instructional practices adjustment and perceived efficacy in classroom management.

The dependent variables of the Facilitators will be collected in three moments: 1) before conducting the EBS Training; 2) at the end of the EBS Training, and 3) at the end of the period of simulations in the subjects Practicum I, III and V of the corresponding courses.

Student variables:

Independent variables:

Sociodemographic data: subject (Practicum I, III, V), age, gender, previous work experience in the health field. These variables will be collected at baseline.

Simulation-based education:

As described above, each student in the Practicum I, III and V subjects will carry out a simulation session based on the context of the subject taken.

The simulations are carried out in groups of 5 students who have the same UVic tutor in common who acts as Facilitator during the simulation. Each simulation is applied following the three previously described phases (prebriefing, simulation per se and debriefing) and the progression between the different subjects places more emphasis on these phases.

Practicum I: the prebriefing has more value in order to guarantee the safety and confidence of the group of students. The simulation per se is developed by two volunteer students. The debriefing is shorter, not very demanding with the result of the case, the objectives are investigated, but without going into excessive depth, undervaluing the error and overvaluing the learning of the students.

Practicum III: the representation of the prebriefing and the debriefing is equalized. The simulation per se is developed by a single volunteer student.

Practicum V: increases the demand of the case, so that it is not necessary to carry out such an extensive prebriefing, but all the parts of the briefing are reviewed, highlighting the objectives to be worked on. The debriefing is more demanding, reflective and complete, with a greater burden of transfer to the real clinical space. The simulation per se is developed by only 1 volunteer student.

Dependent variables:

Dependent variables 1, 2 and 3 of the students will be collected prior to the EBS period in the Practicum I, III and V subjects of the corresponding courses and after the completion of the EBS. Dependent variables 4 and 5 will only be collected after the completion of the EBS period of the corresponding subjects.

All the questionnaires that will be used will be self-administered and will be administered in Spanish.

Perceived self-efficacy specific to academic situations. It will be assessed using the Specific Perceived Self-Efficacy of Academic Situations (AEPESA) scale, which is made up of 10 items that aim to measure self-efficacy expectations in specific situations of the educational context in adolescent and university students.

Academic commitment of university students. It will be assessed using the Well-being in the academic context questionnaire or Utrecht Work Engagement Scale (UWES). It includes the following dimensions:

Academic vigor, measures students' energy, resilience, and willingness to invest effort in their studies.

Academic dedication, assesses students' psychological involvement and commitment to their studies.

Academic absorption, measures students' ability to be completely immersed in their studies.

Satisfaction and confidence regarding EBS, using the Student Satisfaction and Self-Confidence in Learning (SCLC) questionnaire.

Students' perception of the best educational practices in simulation, through the questionnaire on educational practices (EPQ-Sp).

In phase 2, qualitative data will be collected through online focus group interviews, once the EBS and evaluation period of the Physiotherapy Degree students has ended.

A researcher, without a relationship of superiority over the students, will contact the selected students via email and invite them to participate in a single FG.

All FGs will have the same structure: 1) presentation and introduction, in which the participants and the facilitator will introduce themselves; 2) group discussion, in which the facilitator will ask questions based on the script in a flexible way; and 3) conclusions and closure. All FGs will be video and voice recorded to ensure that no data is lost and the researcher will note any relevant aspects observed during the discussions.

Data analysis

Phase 1. Quantitative analysis:

For statistical analysis, the computer program "The Statistical Package for the Social Sciences" will be used. To analyze the distribution of data related to the facilitators, the Shapiro-Wilk test (p> 0.05) will be used, and for student data, the Kolmogorov-Smirnov test (p> 0.05).

In the case of objectives 1.1. and 1.2., descriptive statistics will be used. In the event that the data follow a normal distribution, parametric tests such as the repeated measures ANOVA analysis of variance will be applied to assess the change over time for the study variables. To assess the change in the study variables in the different periods, the Student T-test of related measures will be applied. The Bonferroni correction will be applied for multiple comparisons. In the event that the data do not follow a normal distribution, non-parametric tests such as Friedmann's ANOVA and the Wilcoxon Signed Rank Test will be applied.

For objective 1.3. a descriptive analysis of the study variables will be carried out.

Phase 2. Qualitative analysis:

The data to be analyzed in this case will be the transcriptions of the FG recordings. First, the voice recordings will be transcribed verbatim. The notes taken during the FG will be incorporated as a "commentary." During the transcription process, the identifying information of the participants will be removed and the data will be coded using numerical codes. After coding the files with the same numerical code for each FG, they will be stored on the UVic-UCC Office 365 server. Once coded, the transcripts will be sent to the participants for their approval. If any participant considers making any changes to the transcripts, the interviewer will repeat the data verification process until obtaining their approval of the transcription. Once approved, the voice and video recording files will be deleted.

The entire qualitative analysis process will be carried out using the Atlas.ti software. In the first phase, all transcripts will be read and re-read to familiarise themselves with the data, and primary themes will be generated. In the second phase, the provisional list of primary themes will be organised into groups of "codes". In the third phase, the codes will be applied across all transcripts for analysis.

ELIGIBILITY:
The following inclusion and exclusion criteria have been established for the student population:

Inclusion criteria:

1. First enrollment in the Pràcticum I, III, or V courses.
2. Completion of the full SBE session.

Exclusion criteria:

a) Failure to achieve a grade of 5 in any of the evaluative components of the course.

Regarding the inclusion and exclusion criteria established for the facilitators:

Inclusion criteria:

a) Facilitator of simulations in the Pràcticum I, III, or V courses.

Exclusion criteria:

a) Failure to attend both training sessions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Perceived Self-Efficacy in Academic Situations | Baseline (pre-SBE), 3 months (Post-SBE)
  collected on student population. This will be assessed using the Perceived Self-Efficacy in Academic Situations Scale (AEPESA), which consists of 10 items aimed at measuring self-efficacy expectations in specific educational contexts for adolescent and university students. The 10 items are evaluated using a 10-point Likert scale. The total score reflects the degree of perceived academic self-efficacy, with higher scores indicating greater self-efficacy. This scale has been widely used in psychology studies in university settings.
Behavior to Facilitate Student Learning During SBE | Baseline (pre-capacitation), 3 months (pre-SBE), 4 months (post-SBE)
  collected on facilitator population
  This will be assessed using the Evaluation of Debriefing for Simulation in Healthcare (EDSS). This scale evaluates facilitator behaviors that promote learning and change in experiential contexts by analyzing six key elements of debriefing. These include "if" and "how" the instructor:
  Establishes a stimulating learning environment. Maintains a stimulating learning environment. Structures the debriefing in an organized manner. Provokes stimulating discussions. Identifies and explores performance gaps. Helps students achieve or sustain good performance in the future. The questionnaire consists of 23 items rated on a 7-point Likert scale, where 1 is "extremely ineffective" and 7 is "extremely effective." The EDSS is a behavior-anchored evaluation scale, meaning it is based on behaviors necessary for effective debriefing, as well as those characteristic of ineffective debriefing.

SECONDARY OUTCOMES:
Academic Engagement of University Students | Baseline (pre-SBE), 3 months (Post-SBE)
  collected on student population.
  This will be assessed using the Utrecht Work Engagement Scale, adapted for academic contexts. Originally designed for workplace settings, it has been adapted to evaluate students' engagement in their studies. The scale includes the following dimensions:
  1. Academic Vigor: Measures energy, resilience, and willingness to invest effort in studies.
  2. Academic Dedication: Assesses involvement and psychological commitment to studies.
  3. Academic Absorption: Evaluates the ability to be fully immersed in studies.
  The scale consists of 17 items evaluated on a 6-point Likert scale (1 = "never or almost never," 6 = "always or every day"). Higher scores indicate greater engagement. It has been widely used in psychology studies in academic contexts.
Empathy in Health Science Students | Baseline (pre-SBE), 3 months (Post-SBE)
  collected on student population Empathy will be assessed using the Jefferson Scale of Empathy (JSE), which evaluates the ability to understand and relate to patients' experiences and perspectives. The scale consists of 20 items evaluated on a 7-point Likert scale (1 = "strongly disagree," 7 = "strongly agree"). Higher scores indicate greater empathy. This scale has been widely used in psychology studies in university settings.
Satisfaction and Confidence Regarding SBE | 3 months (Post-SBE)
  collected on student population. This will be measured using the Student Satisfaction and Self-Confidence in Learning Questionnaire (SCLC). The questionnaire consists of 13 items divided into two dimensions: attitudes toward satisfaction with instruction and self-confidence in simulation-based learning. Each item is evaluated using a 5-point Likert scale (1 = "strongly disagree," 5 = "strongly agree"). The total scores for each dimension indicate the levels of satisfaction and self-confidence in clinical simulation learning. Psychometric properties have shown adequate internal consistency and construct validity, with a Cronbach's alpha of 0.885 for the overall questionnaire and >0.81 for each dimension, indicating reliability.
Perception of Educational Best Practices in Simulation | 3 months (Post-SBE)
  collected on student population. This will be assessed using the Educational Practices Questionnaire (EPQ-Sp) (Annex 9), designed to evaluate students' perceptions of educational practices in simulation and their levels of satisfaction and self-confidence. The questionnaire includes 16 items grouped into four dimensions: active learning, collaboration, different learning methods, and expectations. Each item evaluates both the presence and importance of good educational practices in clinical simulation using a 5-point Likert scale (1 = "strongly disagree," 5 = "strongly agree"). Psychometric properties have shown adequate internal consistency and construct validity, with a Cronbach's alpha ≥ 0.70 for the overall questionnaire and each dimension.
Teaching Self-Efficacy Using the Teaching Self-Efficacy Scale | Baseline (pre-capacitation), 3 months (pre-SBE), 4 months (post-SBE)
  collected on facilitator population.
  This will be assessed using the Teaching Self-Efficacy Scale, which consists of 24 items rated on a 5-point Likert scale (from "Not at all" to "To a great extent"). The items are distributed across three dimensions:
  Perceived efficacy in student engagement: Evaluates the teacher's confidence in their ability to positively influence students.
  Perceived efficacy in instructional practices: Assesses the teacher's self-evaluation of their ability to generate alternatives that enhance student performance.
  Perceived efficacy in classroom management: Relates to the teacher's self-evaluation of their ability to maintain classroom order and discipline.

CONTACTS AND LOCATIONS:
Overall Officials: Mirari Ochandorena Acha, doctor, Principal Investigator — UVIC-UCC
Locations (1):
- Universidad de Vic - Universidad Central de Cataluña, Vic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brown L, Ilhan E, Pacey V, Hau W, Van Der Kooi V, Dale M. The Effect of High-Fidelity Simulation-Based Learning in Acute Cardiorespiratory Physical Therapy-A Mixed-Methods Systematic Review. J Phys Ther Educ. junio de 2021;35(2):146-58.
- [Background] Braun V, Clarke V. To saturate or not to saturate? Questioning data saturation as a useful concept for thematic analysis and sample-size rationales. Qual Res Sport Exerc Health. 4 de marzo de 2021;13(2):201-16.
- [Background] Farres-Tarafa M, Bande D, Roldan-Merino J, Hurtado-Pardos B, Biurrun-Garrido A, Molina-Raya L, Raurell-Torreda M, Casas I, Lorenzo-Seva U. Reliability and validity study of the Spanish adaptation of the "Student Satisfaction and Self-Confidence in Learning Scale" (SCLS). PLoS One. 2021 Jul 23;16(7):e0255188. doi: 10.1371/journal.pone.0255188. eCollection 2021. PMID 34297773
- [Background] Dominguez-Lara SA, Fernández-Arata M, Seperak-Viera R. Análisis psicométrico de una medida ultra-breve para el engagement académico: UWES-3S: UWES-3S en estudiantes universitarios. Rev Argent Cienc Comport. 24 de abril de 2021;13(1):25-37.
- [Background] Madsgaard A, Roykenes K, Smith-Strom H, Kvernenes M. The affective component of learning in simulation-based education - facilitators' strategies to establish psychological safety and accommodate nursing students' emotions. BMC Nurs. 2022 Apr 20;21(1):91. doi: 10.1186/s12912-022-00869-3. PMID 35443709
- [Background] Husebo SE, Dieckmann P, Rystedt H, Soreide E, Friberg F. The relationship between facilitators' questions and the level of reflection in postsimulation debriefing. Simul Healthc. 2013 Jun;8(3):135-42. doi: 10.1097/SIH.0b013e31827cbb5c. PMID 23343839
- [Background] Palominos E, Levett-Jones T, Power T, Martinez-Maldonado R. Healthcare students' perceptions and experiences of making errors in simulation: An integrative review. Nurse Educ Today. 2019 Jun;77:32-39. doi: 10.1016/j.nedt.2019.02.013. Epub 2019 Feb 23. PMID 30947020
- [Background] Shoemaker MJ, de Voest M, Booth A, Meny L, Victor J. A virtual patient educational activity to improve interprofessional competencies: A randomized trial. J Interprof Care. 2015;29(4):395-7. doi: 10.3109/13561820.2014.984286. Epub 2014 Nov 21. PMID 25412759
- [Background] King J, Beanlands S, Fiset V, Chartrand L, Clarke S, Findlay T, Morley M, Summers I. Using interprofessional simulation to improve collaborative competences for nursing, physiotherapy, and respiratory therapy students. J Interprof Care. 2016 Sep;30(5):599-605. doi: 10.1080/13561820.2016.1189887. Epub 2016 Jun 24. PMID 27340933
- [Background] Simonson M, Azaiza K, Mitzova-Vladinov G, Bizzio-Knott R, Hooshmand M, Hauglum S, et al. SPECIAL SECTION: TECHNOLOGICAL INNOVATION IN HEALTH CARE EDUCATION. Distance Learn. 14(1).
- [Background] Kolb DA, Boyatzis RE, Mainemelis C. Experiential learning theory: Previous research and new directions. Perspect Think Learn Cogn Styles. 2001;227-47.
- [Background] Hough J, Levan D, Steele M, Kelly K, Dalton M. Simulation-based education improves student self-efficacy in physiotherapy assessment and management of paediatric patients. BMC Med Educ. 2019 Dec 16;19(1):463. doi: 10.1186/s12909-019-1894-2. PMID 31842864